CLINICAL TRIAL: NCT06072248
Title: Effect of Bronchoscopy on the Outcome of Patients With Severe Sepsis With ARDS and Complicated by VAP From Prolonged Ventilation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: icu-23
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: ARDS; Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Meropenem; Bronchoscopy; Ventilators, Mechanical

STUDY DESIGN:
Intervention Model Description: 200 patients included in our study from those who showed no improvement and still had respiratory failure and completed ventilation for 4 days and fulfilled > 2 parameters on SOFA score [9-10] and > 6 on CPIS score and randomly allocated in two groups 100 patients in each.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Placebo Comparator): patients of group A Continue on the conventional way of ventilation and . Microbiological results collected from patients of group A through qualitative sputum.
  Interventions: Drug: Meropenem; Device: ventilator
- Group B (Active Comparator): had three times bronchoscopy one at the end of first 5 days, second bronchoscopy at the end of the second 5 days and last one at the end of the studied period to confirm both clinical and bacteriological cure. Bronchoscopy done with the following precautions: we used flexible bronchoscopy Olympus BF-160 adult size, patients kept sedated with both midazolam and fentanyl, 4 syringe of normal isotonic saline used for wash every one 10 ml and suction done immediately after injection, suction of the fluid and small airway secretion after only the first injection of isotonic saline syringe used for BAL and sent for qualitative culture
  Interventions: Drug: Meropenem; Procedure: bronchoscopy; Device: ventilator

INTERVENTIONS:
Drug: Meropenem — all patients in both groups receive meropenam and put on the ventilators for 2 weeks
Procedure: bronchoscopy — Only patients of group B had three times bronchoscopy according to our protocol one at the end of first 5 days, second bronchoscopy at the end of the second 5 days and last one at the end of the studied period
  Arms: Group B
Device: ventilator — ventilator

SUMMARY:
to evaluate the effect of use of bronchoscopy in the course of sepsis, weaning from the ventilator, duration of ICU stays and mortality rate in septic patients with ARDS due to VAP.

DETAILED DESCRIPTION:
age group between 18-65 years, intubated and ventilated patients due to respiratory failure from severe lung infection and/or traumatic lung contusion [respiratory failure was diagnosed by arterial blood gases (ABG) with partial pressure of oxygen (PaO2) ≤60 mmHg, partial pressure of carbon dioxide (PaCO2)≥60 mmHg, PH > 7.30, respiratory rate >25 min]. All patients ventilated for 4 days with CMV with respiratory rate 12/min, PEEP 5 cm/H2O, FIO2 adjusted to maintain arterial oxygen saturation above 90%. And sedated with both fentanyl and midazolam intravenous infusion to adjust sedation level to achieve Richmond Agitation-Sedation Scale (RASS) -2 to -3 as illustrated in table. All patients received broad spectrum antibiotics in form of meropenem 1 gm slowly intravenous every 8 hours in this period (four days) and a qualitative sputum culture collected from all patients after 3 days from ventilation. Feeding started on the second day of ventilation to all patients through feeding pump at rate of 70 ml insure plus (Abbot company) with 1.47 kilo-calorie/ml to supply patients with approximately 2500 kilo-calorie in 24 hours calculated by approximately 35 kilo-calorie/kg. The 5 points of bundle for pneumonia prevention were strictly applied to all patients: Elevation of the head of the bed 30º to 45º, Daily evaluation for possible ex-tubation, The use of endotracheal tube with subglottic secretion drainage, oral care with oral antiseptics, initiation of safe enteral nutrition, within 24-48 hours from ICU admission and ventilation.

200 patients included in our study from those who showed no improvement and still had respiratory failure and completed ventilation for 4 days and fulfilled > 2 parameters on SOFA score and > 6 on pneumonia score and randomly allocated in two groups 100 patients in each. Randomization sequence was created using Excel 2007 (Microsoft, Redmond, WA, USA) with a 1:1 allocation using random block sizes of 2 and 4 by an independent doctor. In this way, sequence generation and type of randomization can be expressed at the same time.

All patients selected underwent a percutaneous tracheostomy on the same day. Sepsis documented in our study by > 2 on Sequential Organ Failure Assessment (SOFA) score. While VAP documented in our study by >6 on CPIS score. Only patients of group B had three times bronchoscopy according to our protocol one at the end of first 5 days, second bronchoscopy at the end of the second 5 days and last one at the end of the studied period to confirm both clinical and bacteriological cure. Bronchoscopy done with the following precautions: we used flexible bronchoscopy Olympus BF-160 adult size, patients kept sedated with both midazolam and fentanyl infusion to get same sedation score mentioned before (RASS-2/-3), increase FIO2 to 100% during the procedure, use xylocaine spray 10% by Astra Zeneca company 2 puffs in each nostril before application of the rubber tube of the bronchoscope, keep patient's head elevated 20 degree during procedure, use CMV mode with previous mentioned parameters with 100% FIO2 during the procedure, 4 syringe of normal isotonic saline used for wash every one 10 ml and suction done immediately after injection, suction of the fluid and small airway secretion after only the first injection of isotonic saline syringe used for BAL and sent for qualitative culture and the other isotonic saline injected in the remaining three syringe used only for wash the small airways and not for bacteriological sampling, monitoring of patients during the procedure done by SPO2, non-invasive blood pressure measurement every 5 minutes, electro cardiac gram for heart rate, clinical assessment of depth of sedation every 5 minutes.

Duration of the study selected to be 2 weeks and evaluation of all patients in both groups done on three periods, at the end of the first 5 days, at the end of the second 5 days and at the end of last 4 days.

ELIGIBILITY:
Inclusion Criteria:

* patients with age group between 18-65 years,patients Respiratory failure, patients with pneumonia

Exclusion Criteria:

* pediatric patients, patients with anoxic brain insult

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only adult patients from both sexes
Enrollment: 200 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
number of patients weaned from the ventilator | 2 weeks
  those who had improvement in all parameters of sepsis (SOFA score) and improvement in (CPIS) score
number of patients disharged from ICU | 2 weeks
  Those who weaned from the ventilator and recoverd from sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No